CLINICAL TRIAL: NCT05874505
Title: "Multicenter, Randomized, Prospective Trial Comparing the Efficacy and Safety of Adalimumab to That of Tocilizumab in Severe Uveitis of Behçet's Disease" (UVB) : Treatment of UVeitis in Behçet's Diseases With Biologics
Brief Title: "Comparison of the Efficacy and Safety of Adalimumab to That of Tocilizumab in Severe Uveitis of Behçet's Disease"
Acronym: UVB
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200007
Record Dates: First submitted 2023-04-14; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Behcet's Uveitis
Keywords: Biologics; Adalimumab; Tocilizumab
MeSH Terms: interventions — Adalimumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab (Experimental): Adalimumab 80 mg at Day 0 then 40 mg subcutaneous at week 1, 3, 5, 7, 9, 11, 13 and 15
  Interventions: Drug: Adalimumab
- Tocilizumab (Experimental): Tocilizumab 162 mg subcutaneous each week for 15 weeks
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab 80 mg at Day 0 then 40 mg subcutaneous at week 1, 3, 5, 7, 9, 11, 13 and 15
  Arms: Adalimumab
Drug: Tocilizumab — Tocilizumab 162 mg subcutaneous each week for 15 weeks
  Arms: Tocilizumab

SUMMARY:
UVB, is the first randomized prospective, head to head study, comparing Adalimumab to Tocilizumab in sight threatening uveitis of Behçet's Disease (BD). Anti-TNFα has been used for BD uveitis for 15 years. The incidence of blindness in BD has been dramatically reduced in the recent years with the use of biologics. There is no firm evidence or randomized controlled trials directly addressing the best induction therapy in severe BD uveitis. BD uveitis is considered as the most devastating inflammatory ocular disease. Risk of visual loss reaches 25% at 5 years and 80% of patients have a bilateral involvement. Contrasting with immunosuppressors or interferon-alpha, biotherapies act rapidly and are highly effective in steroid's sparing thus preventing occurrence of cataract and/or glaucoma. However, anti-TNFα failed to demonstrate sustainable complete remission over 50 % of severe sight threatening uveitis. There is little published information on use of biologics other than anti-TNFα for severe BD uveitis. Tocilizumab has been used with success in severe and/or resistant cases and is one of the most promising biologics in BD. IL-6 expression correlates with BD activity and other immunological data provide a strong rationale for targeting BD with tocilizumab. Despite a strong rationale, these compounds are not yet approved in BD, which guarantees the innovative nature of this study that aims selecting or dropping any arm when evidence of efficacy already exists. The objective of the study is to assess the benefit of tocilizumab comparatively to that of adalimumab in sight-threatening Behçet's disease uveitis at week 16

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 at Inclusion
2. Provide written, informed consent prior to the performance of any study-specific procedures
3. Diagnosis of Behçet's disease according to the International Criteria for Behçet's Disease (ICBD) or history of aphthosis.
4. Diagnosis of non-infectious intermediate, posterior-, or pan-uveitis in at least one eye fulfilling the International Study Group Classification Criteria (Standardization of Uveitis Nomenclature [SUN] criteria) of posterior, or pan- uveitis
5. Sight threatening uveitis defined according to the validated international definition as 2 lines of drop in visual acuity on a 10/10 scale, and/or retinal inflammation (macular oedema and/or retinal vasculitis).
6. Chest X-ray (postero-anterior and lateral) or CT-scanner results within 12 weeks prior to Inclusion with no evidence of active Tuberculosis, active infection, or malignancy
7. For female subjects of childbearing potential (premenopausal female capable of becoming pregnant) , a negative serum pregnancy test (plasmatic or urinary)
8. For subjects with reproductive potential, a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study and 3 and 5 months after stopping therapy for tocilizumab and adalimumab, respectively. Birth control methods which may be considered as highly effective methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods (according to CTFG recommendations). Such methods include:

   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * oral
     * intravaginal
     * transdermal
   * progestogen-only hormonal contraception associated with inhibition of ovulation:

     * oral
     * injectable
     * implantable
   * intrauterine device (IUD)
   * intrauterine hormone-releasing system (IUS)
   * bilateral tubal occlusion
   * vasectomised partner
   * sexual abstinence (In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject).

   For male subjects :
   * use of a condom
   * vasectomy (with documentation of azoospermia)
   * sexual abstinence
9. A potential subject with a positive interferon-gamma release assay (IGRA) (e.g., QuantiFERON®-TB Gold or T-spot TB® Test) obtained within 6 months prior to inclusion is eligible if her/his chest X-ray does not show evidence suggestive of active TB disease and there are no clinical signs and symptoms of pulmonary and/or extra-pulmonary TB disease. These subjects with a latent TB infection who have not already received a prophylactic TB treatment must agree in advance to complete such a treatment course. The treatment should be started at the latest at inclusion.
10. Affiliation to a social security system. Patients affiliated to universal medical coverage (CMU) are eligible for the study

Exclusion Criteria:

1. Infectious uveitis, masquerade syndromes, or uveitis due to causes other than BD uveitis
2. Active tuberculosis or history of untreated tuberculosis and/or severe infection
3. Positive HIV antibody and/or positive hepatitis B surface antigen and/or positive hepatitis C RNA, results obtained within 1 month prior to inclusion
4. History of malignancy within 5 years prior to Inclusion other than carcinoma in situ of the cervix or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin.
5. History of severe allergic or anaphylactic reactions to monoclonal antibodies
6. History of multiple sclerosis and/or demyelinating disorder
7. Hypersensitivity to the active substance or an excipient of the Investigational Medicinal Product or the auxiliary medicine
8. Active or suspected ocular infection
9. Active or suspected systemic infection
10. History of intestinal ulceration or diverticulitis
11. Known porphyria
12. Laboratory values assessed during Inclusion:

    1. Neutrophil < 1.0 x 10^3 /mm3
    2. Platelet count < 80 x 10^3 /mm3
    3. ASAT or ALAT > 5 ULN
13. Treatment with anti-TNF and/or Tocilizumab therapy within 1 month prior to inclusion
14. if on azathioprine, mycophenolate mofetil, or methotrexate at the time of inclusion, these drugs must be withdrawn prior to receiving the tocilizumab or adalimumab dose on Day 0
15. Stage III and IV New York Heart Association (NYHA) cardiac insufficiency
16. Severe renal (Glomerular filtration rates (GFR) <30ml/min) or liver insufficiency (prothrombin <50% without other causes)
17. Any live (attenuated) vaccine within 4 weeks prior to inclusion
18. Breastfeeding or pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete remission of ocular involvement (Efficacy) | At week 16 after randomization
  Efficacy will be defined by a complete remission of ocular involvement with prednisone lower or equal to 5 mg/day . Ocular involvement response to treatment will be evaluated according to the Standardization of Uveitis Nomenclature (SUN) Workgroup criteria.

SECONDARY OUTCOMES:
Percent of patients meeting the corticosteroid sparing targets | At week 16 after randomization
  lower than 0.1 mg/day/kg of prednisone
Mean dose of corticosteroids | At week 16 after randomization
Cumulative dose of corticosteroids | At week 16 after randomization
Time to response onset | Up to week 48
Erythrocyte sedimentation rate | At week 4
Erythrocyte sedimentation rate | At week 8
Erythrocyte sedimentation rate | At week 12
Erythrocyte sedimentation rate | At week 16
Erythrocyte sedimentation rate | At week 24
Erythrocyte sedimentation rate | At week 36
Erythrocyte sedimentation rate | At week 48
C-reactive protein rate | At week 4
C-reactive protein rate | At week 8
C-reactive protein rate | At week 12
C-reactive protein rate | At week 16
C-reactive protein rate | At week 24
C-reactive protein rate | At week 36
C-reactive protein rate | At week 48
Rate of relapses | up to 48 weeks
  Relapse will be defined as the reappearance of clinical and/or paraclinical features of active disease or by the occurrence of new lesions or progression of preexisting lesions
Time to occurrence of relapse or worsening of uveitis | up to 48 weeks
  Relapse will be defined as the reappearance of clinical and/or paraclinical features of active disease or by the occurrence of new lesions or progression of preexisting lesions
Disease activity assessed by Behcet's Disease Current Activity | At week 8
  Changes in Behcet's Disease Current Activity Form 2006 The score varies between 0 and 12, the higher the score the higher the disease activity.
  Lawton G, Bhakta BB, Chamberlain MA, Tennant A. The Behcet's disease activity index. Rheumatology (Oxford). 2004 Jan;43(1):73-8. doi: 10.1093/rheumatology/keg453. Epub 2003 Jul 30. PMID: 12890862.
Disease activity assessed by Behcet's Disease Current Activity | At week 16
  Changes in Behcet's Disease Current Activity Form 2006 The score varies between 0 and 12, the higher the score the higher the disease activity.
  Lawton G, Bhakta BB, Chamberlain MA, Tennant A. The Behcet's disease activity index. Rheumatology (Oxford). 2004 Jan;43(1):73-8. doi: 10.1093/rheumatology/keg453. Epub 2003 Jul 30. PMID: 12890862.
Disease activity assessed by Behcet's Disease Current Activity | At week 24
  Changes in Behcet's Disease Current Activity Form 2006 The score varies between 0 and 12, the higher the score the higher the disease activity.
  Lawton G, Bhakta BB, Chamberlain MA, Tennant A. The Behcet's disease activity index. Rheumatology (Oxford). 2004 Jan;43(1):73-8. doi: 10.1093/rheumatology/keg453. Epub 2003 Jul 30. PMID: 12890862.
Disease activity assessed by Behcet's Syndrome Activity Score | At week 8
  Changes in Behcet's Syndrome Activity Score. It is a 10 items score. The score varies between 0 and 100. The higher the score the higher the disease activity.
  Forbees C, Swearingen C, Yazici Y. Behcet's syndrome activity score (BSAS): a new disease activity assessment tool, composed of patient-derived measures only, is strongly correlated with the Behcet's Disease Current Activity Form (BDCAF) Arthritis Rheum. 2008;58(Suppl 9):S854-S855.
Disease activity assessed by Behcet's Syndrome Activity Score | At week 16
  Changes in Behcet's Syndrome Activity Score. It is a 10 items score. The score varies between 0 and 100. The higher the score the higher the disease activity.
  Forbees C, Swearingen C, Yazici Y. Behcet's syndrome activity score (BSAS): a new disease activity assessment tool, composed of patient-derived measures only, is strongly correlated with the Behcet's Disease Current Activity Form (BDCAF) Arthritis Rheum. 2008;58(Suppl 9):S854-S855.
Disease activity assessed by Behcet's Syndrome Activity Score | week 24
  Changes in Behcet's Syndrome Activity Score It is a 10 items score. The score varies between 0 and 100. The higher the score the higher the disease activity.
  Forbees C, Swearingen C, Yazici Y. Behcet's syndrome activity score (BSAS): a new disease activity assessment tool, composed of patient-derived measures only, is strongly correlated with the Behcet's Disease Current Activity Form (BDCAF) Arthritis Rheum. 2008;58(Suppl 9):S854-S855.
Changes in the number of other organs involved by Behcet Disease (BD) | At week 4
Changes in the number of other organs involved by Behcet Disease (BD) | At week 8
Changes in the number of other organs involved by Behcet Disease (BD) | At week 12
Changes in the number of other organs involved by Behcet Disease (BD) | At week 16
Changes in the number of other organs involved by Behcet Disease (BD) | At week 24
Changes in the number of other organs involved by Behcet Disease (BD) | At week 36
Changes in the number of other organs involved by Behcet Disease (BD) | At week 48
Quality of Life assessed by Behcet's Disease Quality of Life Measure | At week 16
  It is a score composed of 30 items and the result varies between 0 and 30. The higher the score, the lower the quality of life.
  G. Gilworth, MA Chamberlain, B. Bhakta, A. Silman, D. Haskard and A. Tennant. (2004), The Development of the BD-Qol: A Quality of Life Instrument Specific to Behçet's Disease., J Rheum, 31, 931-7
Quality of Life assessed by Behcet's Disease Quality of Life Measure | At week 24
  It is a score composed of 30 items and the result varies between 0 and 30. The higher the score, the lower the quality of life.
  G. Gilworth, MA Chamberlain, B. Bhakta, A. Silman, D. Haskard and A. Tennant. (2004), The Development of the BD-Qol: A Quality of Life Instrument Specific to Behçet's Disease., J Rheum, 31, 931-7
Changes in Short Form (36) Health Survey for quality of life | At week 16
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
  Ware JE, Sherbourne CD. The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Med Care 1992;30:473-83.
Changes in Short Form (36) Health Survey for quality of life | At week 24
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
  Ware JE, Sherbourne CD. The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Med Care 1992;30:473-83.
Proportion of patients with adverse clinical events | at week 4
Proportion of patients with adverse clinical events | at week 8
Proportion of patients with adverse clinical events | at week 12
Proportion of patients with adverse clinical events | at week 16
Proportion of patients with adverse clinical events | at week 24
Proportion of patients with adverse clinical events | at week 36
Proportion of patients with adverse clinical events | at week 48
Severity of adverse clinical events | At week 4
  It is determined according to the Common Terminology Criteria for Adverse Events (CTCAE). The grade varies from 1 to 5. Grade 1 corresponds to mild severity and grade 5 to death.
Severity of adverse clinical events | At week 8
  It is determined according to the Common Terminology Criteria for Adverse Events (CTCAE). The grade varies from 1 to 5. Grade 1 corresponds to mild severity and grade 5 to death. death.
Severity of adverse clinical events | At week 12
  It is determined according to the Common Terminology Criteria for Adverse Events (CTCAE). The grade varies from 1 to 5. Grade 1 corresponds to mild severity and grade 5 to death.
Severity of adverse clinical events | At week 16
  It is determined according to the Common Terminology Criteria for Adverse Events (CTCAE). The grade varies from 1 to 5. Grade 1 corresponds to mild severity and grade 5 to death.
Severity of adverse clinical events | At week 24
  It is determined according to the Common Terminology Criteria for Adverse Events (CTCAE). The grade varies from 1 to 5. Grade 1 corresponds to mild severity and grade 5 to death.
Severity of adverse clinical events | At week 36
  It is determined according to the Common Terminology Criteria for Adverse Events (CTCAE). The grade varies from 1 to 5. Grade 1 corresponds to mild severity and grade 5 to death.
Severity of adverse clinical events | At week 48
  It is determined according to the Common Terminology Criteria for Adverse Events (CTCAE). The grade varies from 1 to 5. Grade 1 corresponds to mild severity and grade 5 to death.
Changes in Tyndall score | At week 8
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to grade 4+. The higher the grade the higher the number of cells in the anterior chamber.
Changes in Tyndall score | At week 16
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to grade 4+. The higher the grade the higher the number of cells in the anterio chamber.
Changes in Tyndall score | At week 24
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to grade 4+. The higher the grade the higher the number of cells in the anterior chamber.
Changes in Tyndall score | At week 36
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to grade 4+. The higher the grade the higher the number of cells in the anterior chamber.
Changes in Tyndall score | At week 48
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to grade 4+. The higher the grade the higher the number of cells in the anterior chamber.
Changes in flare score | At week 8
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to 4+. The higher the score, the higher the inflammation.
Changes in flare score | At week 16
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to 4+. The higher the score, the higher the inflammation.
Changes in flare score | At week 24
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to 4+. The higher the score, the higher the inflammation.
Changes in flare score | At week 36
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to 4+. The higher the score, the higher the inflammation.
Changes in flare score | At week 48
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies from grade 0 to 4+. The higher the score, the higher the inflammation.
Changes of Vitreous Haze | At week 8
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies between 0 and 4. The higher the score the higher the inflammation.
Changes of Vitreous Haze | At week 16
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies between 0 and 4. The higher the score the higher the inflammation.
Changes of Vitreous Haze | At week 24
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies between 0 and 4. The higher the score the higher the inflammation.
Changes of Vitreous Haze | At week 36
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies between 0 and 4. The higher the score the higher the inflammation.
Changes of Vitreous Haze | At week 48
  The score is calculated according to the Standardization of Uveitis Nomenclature (SUN). It varies between 0 and 4. The higher the score the higher the inflammation.
Changes in Best corrected visual acuity | At week 8
  Evaluated by Early Treatment Diabetic Retinopathy Study (ETDRS) letters score. The total score varies between 0 and 100. The higher score the better the visual acuity.
  ETDRS Early Treatment Diabetic Retinopathy Study Research Group Treatment Diabetic Retinopathy Study design and baseline patient characteristics. ETDRS report number 7., Ophthalmology. 1991 May; 98(5 Suppl):741-756
Changes in Best corrected visual acuity | At week 16
  Evaluated by ETDRS letters score. The total score varies between 0 and 100. The higher score the better the visual acuity
  ETDRS Early Treatment Diabetic Retinopathy Study Research Group Treatment Diabetic Retinopathy Study design and baseline patient characteristics. ETDRS report number 7., Ophthalmology. 1991 May; 98(5 Suppl):741-756
Changes in Best corrected visual acuity | At week 24
  Evaluated by ETDRS letters score. The total score varies between 0 and 100. The higher score the better the visual acuity
  ETDRS Early Treatment Diabetic Retinopathy Study Research Group Treatment Diabetic Retinopathy Study design and baseline patient characteristics. ETDRS report number 7., Ophthalmology. 1991 May; 98(5 Suppl):741-756
Changes in Best corrected visual acuity | At week 36
  Evaluated by ETDRS letters score. The total score varies between 0 and 100. The higher score the better the visual acuity
  ETDRS Early Treatment Diabetic Retinopathy Study Research Group Treatment Diabetic Retinopathy Study design and baseline patient characteristics. ETDRS report number 7., Ophthalmology. 1991 May; 98(5 Suppl):741-756
Changes in Best corrected visual acuity | At week 48
  Evaluated by ETDRS letters score. The total score varies between 0 and 100. The higher score the better the visual acuity
  ETDRS Early Treatment Diabetic Retinopathy Study Research Group Treatment Diabetic Retinopathy Study design and baseline patient characteristics. ETDRS report number 7., Ophthalmology. 1991 May; 98(5 Suppl):741-756
Changes in central retinal thickness | At week 8
  Changes in central retinal thickness measured with Optical Coherence Tomography (OCT)
Changes in central retinal thickness | At week 16
  Changes in central retinal thickness measured with Optical Coherence Tomography (OCT)
Changes in central retinal thickness | At week 24
  Changes in central retinal thickness measured with Optical Coherence Tomography (OCT)
Changes in central retinal thickness | At week 36
  Changes in central retinal thickness measured with Optical Coherence Tomography (OCT)
Changes in central retinal thickness | At week 48
  Changes in central retinal thickness measured with Optical Coherence Tomography (OCT)
Percentage of patients with central retinal thickness <300 microns | At week 8
Percentage of patients with central retinal thickness <300 microns | At week 16
Percentage of patients with central retinal thickness <300 microns | At week 24
Percentage of patients with central retinal thickness <300 microns | At week 36
Percentage of patients with central retinal thickness <300 microns | At week 48
Percentage of patients without retinal vessel leakage on retinal angiography | At week 16
  in case of retinal vasculitis
Percentage of patients without retinal vessel leakage on retinal angiography | At week 24
  in case of retinal vasculitis
Percentage of patients without retinal vessel leakage on retinal angiography | At week 36
  in case of retinal vasculitis
Percentage of patients without retinal vessel leakage on retinal angiography | At week 48
  in case of retinal vasculitis

IPD SHARING:
Plan to Share IPD: Undecided